CLINICAL TRIAL: NCT04820361
Title: Effect of Cannabinoids on Pain in Fabry Disease Patients; a Prospective, Randomized, Double-blind, Placebo-controlled, Crossover, Multicenter Study
Brief Title: Effect of Cannabinoids on Pain in Fabry Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albina Nowak, MD (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Albina Nowak, MD, Sponsorl Investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Cannabinoids in Fabry pain
Record Dates: First submitted 2020-12-08; First posted 2021-03-29 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pain, Neuropathic
MeSH Terms: conditions — Neuralgia | interventions — Parasympatholytics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: PROSPECTIVE, RANDOMIZED, DOUBLE-BLIND, PLACEBO- CONTROLLED, CROSSOVER, MULTICENTER STUDY.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): oral spray
  Interventions: Drug: Placebo
- Sativex® (Active Comparator): .It contains Δ-9-Tetrahydrocannabinol (THC) and Cannabidiol (CBD)
  Interventions: Drug: Cannabis sativa L., folium cum flore

INTERVENTIONS:
Drug: Cannabis sativa L., folium cum flore — Muscle Relaxation
  Other Names: Spasmolytic
  Arms: Sativex®
Drug: Placebo — Muscle Relaxation
  Other Names: Spasmolytic
  Arms: Placebo

SUMMARY:
Fabry Disease (FD) is a rare lysosomal storage disorder due to the absence or deficiency of hydrolase α-galactosidase A (α-Gal A) activity in lysosomes. This dysfunction results in progressive accumulation of glycosphingolipids in a wide variety of cells, resulting in major organ system damage.

Patients with Fabry disease can suffer from neuropathic pain, since lysosomal accumulation affects small unmyelinated nerve fibers. Neuropathic pain is one of the prominent and debilitating symptoms significantly interfering with life quality in FD patients. Current treatment of Fabry patients with neuropathic pain is deficient, as they respond poorly to a conventional pain therapy, often require a high-dose opioids treatment and presentation to the Emergency Department.

Sativex® has been shown to be a successful treatment option in neuropathic pain of different origin with minimal neuropsychological influence: in multiple sclerosis (MS), chemotherapy-induced neuropathic pain and other. It contains Δ-9-Tetrahydrocannabinol (THC) and Cannabidiol (CBD) and has recently been licensed in Switzerland for treatment of neuropathic chronic pain in MS. Sativex® is an oral spray.

DETAILED DESCRIPTION:
Fabry disease is an X-linked lysosomal storage disease caused by a deficiency of the enzyme α-galactosidase A. Patients suffering from Fabry's disease may suffer from neuropathic pain, since the lysosomal accumulation of lipids can also take place in the small nerve fibers. Typically, neuropathic pain occurs in late childhood or adolescence and disappears after several years, probably due to the irreversible destruction of the small nerve fibers. The pain management of Fabry patients suffering from neuropathic pain is inadequate, as patients often do not respond well to conventional pain therapies.

Aim of this study:

The aim of this study is to find out how strongly the investigational drug Sativex® (active ingredients: tetrahydrocannabinol (THC) and cannabidiol (CBD)) can influence the pain that can be caused by Fabry's disease. For this purpose, the investigational drug is compared with a placebo drug. The latter is a drug without an active ingredient. These studies provide us with important information on the origin of the pain and at the same time on the mechanism of action of Sativex®. This makes it possible to develop new forms of therapy in the future.

Procedure:

A total of 22-30 patients are divided into two groups of 11-15 patients each. Both groups will undergo the same test program. This will be divided into two phases: In the first phase, which will last 8 weeks, one group will receive Sativex® while the other group will receive a placebo. In the second phase, which will also last 8 weeks, the group that previously received the investigational drug will now receive the placebo and the previous placebo group will now receive the investigational drug. The study is double-blind, i.e. neither the patient nor the investigator knows who is receiving the investigational drug or the placebo. Patients are randomly assigned to the groups. Throughout the treatment, patients maintain their usual pain management regimen. (see Study Schedule) For 14 weeks, patients will fill out their pain diary daily. Every two weeks a blood sample is taken to determine the levels of cannabinoid metabolites. At the beginning, at the end of the first and after the second phase, the patient will fill out various questionnaires on neuropathic pain and improvement of quality of life. This will be used to assess whether pain relief is achieved.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* • Age: 18-70 years

  * Patients with genetically confirmed Fabry disease
  * On treatment with Enzyme Replacement Therapy (ERT)
  * Sufficient command of German language
  * Pain duration of more than 3 months
  * Stable analgesic regimen for at least 2 weeks preceding the study entry day
  * Baseline worst last week pain intensity ≥4 on numerical rating scale (NRS)
  * Signed and dated informed consent
  * ERT or chaperone therapy at a stable dose for at least 3 last months

Exclusion Criteria:

* • Known hypersensitivity or allergy to cannabinoids.

  * Women who are pregnant or breast feeding; intention to become pregnant during the course of the study, lack of safe contraception, defined as: female subjects of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not willing or able to use any other second (additional) considered sufficiently reliable by the investigator in individual cases. Female subjects who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
  * Dementia
  * Other pain not of neuropathic origin thought by the investigator to be of nature or severity to interfere with the patient's assessment of neuropathic pain due to Fabry disease.
  * Patients with known or suspected non-compliance, drug or alcohol abuse, including Marijuana cigarettes.
  * Patients with known schizophrenia, other psychotic disorders, personality disorders or another severe psychiatric disorder or positive family history with these disorders, except depression.
  * Patients with another clinically significant disease (e.g. renal failure, hepatic dysfunction, severe cardiovascular or convulsive diseases).
  * Participation in another study with investigational drugs within the 30 days preceding and during the present study.
  * Previous enrolment into the current study
  * Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
NRS | Daily NRS score after 28 days will be compared to baseline NRS score, evaluated before titration phase starts
  NRS is a straightforward commonly used method to illustrate pain.

SECONDARY OUTCOMES:
QST | At baseline and after 28 days of treatment with study drug and placebo, respectively.
  Pain thresholds using the quantitative sensory testing.
WHO-Quality of life score (WHOQOL-BREF) | Between baseline and treatment after 28 days.
  Improvement of quality of life.
Patient global impression of change (PGIC) | For the average pain of treatment week 4.
  Improvement of quality of life.
Short form McGrill Paint Questionnaire (SF-MPQ) | Compared between baseline and average pain of treatment after 28 days.
  Improvement of neuropathic pain.
Douleur Neuropathic en 4 questions (DN4-Questionnaire) | Compared between baseline and treatment week 4.
  Improvement of neuropathic pain.
Profile of Mood States (POMS questionnaire) | Between baseline and treatment week 4.
  Change in Profile of Mood States.
Insomnia severity Index | Between baseline and treatment after 28 days.
  Change in Insomnia severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Albina A Nowak, PH, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zürich USZ, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jensen TS, Baron R. Translation of symptoms and signs into mechanisms in neuropathic pain. Pain. 2003 Mar;102(1-2):1-8. doi: 10.1016/s0304-3959(03)00006-x. No abstract available. PMID 12620591
- [Result] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Result] Serpell M, Ratcliffe S, Hovorka J, Schofield M, Taylor L, Lauder H, Ehler E. A double-blind, randomized, placebo-controlled, parallel group study of THC/CBD spray in peripheral neuropathic pain treatment. Eur J Pain. 2014 Aug;18(7):999-1012. doi: 10.1002/j.1532-2149.2013.00445.x. Epub 2014 Jan 13. PMID 24420962